CLINICAL TRIAL: NCT04650113
Title: Clinical and Radiographic Assessment of Partial and Complete Pulpotomy in Primary Molars Using MTA : A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Assessment of Partial and Complete Pulpotomy in Primary Molars Using MTA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, fatma zainalabdieen abdelraouf, Master degree student, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARopacpIPMUM
Record Dates: First submitted 2020-11-18; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants will be randomly assigned to know which one of the right or left side will be allocated randomly in either the control or the intervention group.
  Sequence Generation Eligible consented participants will be randomly assigned to know which one of the participants will be control or intervention group according to a sequence generated on a Microsoft Excel sheet where the intervention (I) and the control (C) are simply randomized. The table of sequence generation will be kept with the co-supervisor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group A (Experimental): placed with light pressure over the pulpal stumps (if hemorrhage control will not be achieve, tooth will be exclude ) 9.The pellet will be remove, and the pulp chamber filled with MTA. 10.The tooth will prepare and restore with a stainless steel crown cemented with glass ionomer cement
  Interventions: Combination Product: MTA material
- group B (Active Comparator): 1. Pre-operative radiograph showing all roots and their apices.
  2. Local anesthesia will be administered and a rubber dam will take place ,that ensure good isolation of the treated teeth.
  3. Removal of caries
  4. Pulp chambers will access using a no.330 bur in a high-speed hand piece with water coolant.
  5. Removal of any remains of coronal pulp tissue with sharp sterile excavator or large bur in slow hand piece
  6. Pulp amputation will perform using a spoon excavator.
  7. Hemorrhage control will obtain within 5 minutes using sterile cotton pellets placed with light pressure over the pulpal stumps (if hemorrhage control will not be achieve, tooth will be exclude )
  8. The pellet will be remove, and the pulp chamber will be filled with MTA.
  9. The tooth will prepare and restore with a stainless steel crown cemented with glass ionomer cement.
  The periapical radiographic will be taken at this baseline visit .
  Interventions: Combination Product: MTA material

INTERVENTIONS:
Combination Product: MTA material — Partial pulpotomy is a procedure in which the inflamed tissue beneath an exposure is removed to a depth of 1 to 3 mm or deeper to reach healthy pulp tissue.
  Other Names: partial pulpotomy procedure

SUMMARY:
that's comparison between partial and complete pulpotomy techniques in primary teeth

ELIGIBILITY:
Inclusion Criteria:

1. - Medically free children who will be able and cooperative in all steps of the study.
2. - Asymptomatic primary molars with a deep carious lesion.
3. - Vital pulp due to dental caries with no clinical sign of pulpal degeneration (spontaneous pain, fistula, mobility) prior to treatment.

3 - Preliminary radiographs indicating absence of pathologic internal or external root resorption, or any evidence of inter-radicular bone destruction.

4 - Absence of pre-operative pain or they will only have a short-term pain. 5 - No tenderness to percussion. 6-Age ranging 4-6 years.

Exclusion Criteria:

1- Excessive bleeding during pulp amputation. 2 - Non vital teeth. 3 -History of spontaneous or prolonged pain. 4 - Swelling, tenderness, to percussion or palpation, or pathologic mobility. 5 - pre-operative radiographic pathology such as resorption (internal, external); periradicular or furcation radiolucency, or a widened periodontal ligament space.

6 - Parent or guardians who refuse participating in the study

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2021-01-20 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-03 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 1 week
  analog scale
postoperative pain | 1 month
  analog scale
postoperative pain | 3 months
  analog scale
postoperative pain | 6 months
  analog scale
swelling | 1 week
  clinical examination
swelling | 1 month
  clinical examination
swelling | 3 months
  clinical examination
swelling | 6 months
  clinical examination
mobility | 1 week
  clinical examination
mobility | 1 month
  clinical examination
mobility | 3 months
  clinical examination
mobility | 6 months
  clinical examination

SECONDARY OUTCOMES:
root resorption | 1 week
  periapical radiograph
root resorption | 1 month
  periapical radiograph
root resorption | 3 months
  periapical radiograph
root resorption | 6 months
  periapical radiograph
Bone resorption | 1 week
  periapical radiograph
Bone resorption | 1 month
  periapical radiograph
Bone resorption | 3 months
  periapical radiograph
Bone resorption | 6 months
  periapical radiograph

CONTACTS AND LOCATIONS:
Overall Officials: adel El-bardissy, prof, Study Director — Associate Professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry cairo university; rasha ragab, phd, Study Director — Lecturer of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry cairo university
Locations (1):
- Faculty of dentistry cairo university, Al Manyal, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided